CLINICAL TRIAL: NCT06469320
Title: Urinary Incontinence and Other Pelvic Floor Dysfunctions in Trail Runners: Epidemiology and Identification of Risk Factors
Brief Title: Urinary Incontinence and Other Pelvic Floor Dysfunctions in Trail Runners
Acronym: IU-TRAIL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/CHU/13
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online questionnaire — Pelvic floor dysfunction assessment questionnaire adapted from PFD-Sentinel

SUMMARY:
The pelvic floor is a crucial complex for many bodily functions, supporting the pelvic organs and contributing to urinary and anal continence, as well as sexual function. Dysfunction of this structure can lead to a variety of disorders, including urinary incontinence (UI), a common problem in women. Although the prevalence of UI in middle-aged women has been documented at between 20% and 30%, high-impact physical activities, such as certain sports and running, increase the risk of UI. According to the most recently published meta-analysis, the prevalence is 44% [95%CI 30.2-57.8]. Although this subject is often taboo, it can have psychosocial consequences and affect sporting activities. Only 31.7% of female runners talk to a health professional about it. Trail running, a fast-growing discipline, differs from road running in its particular physical demands, which could influence the occurrence of pelvic floor disorders (PFD) and exercise-induced UTIs. The unique characteristics of trail running, such as the technical nature of the terrain, the steep gradients and the variety of distances, place intense demands on the female pelvi-perineal system. Nevertheless, despite the growing popularity of this sport, little epidemiological data exists on the prevalence of stress UTI and pelvic floor disorders among female trail runners.

ELIGIBILITY:
Inclusion Criteria:

* Adult runner
* Residing in mainland France, or in French overseas departments and territories such as Guadeloupe, Martinique, French Guiana, Réunion, Mayotte and New Caledonia
* Practising trail running on a regular basis (defined pragmatically by the participant herself), whether or not affiliated to a club
* Able to complete the questionnaire online-

Exclusion Criteria:

* Pregnant or have given birth in the last six months
* Does not understand French
* A protected adult (guardianship or curatorship) or under court protection

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult french woman practising trail-running
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stress urinary incontinence (SUI) and pelvic floor dysfunction (PFD) | 6 months
  The prevalence will be determined by determining the proportion of female trail runners reporting Stress urinary incontinence and/or Pelvic floor muscle dysfunction out of the total population of trail runners who responded to the questionnaire.

SECONDARY OUTCOMES:
Identify the risk factors associated with SUI and PFD in French trail runners. | 6 months
  Identification of the relative risks of the various suspected risk factors using a multiple logistic regression model
To assess the impact of SUI and PFD on the sporting activities and daily lives of French trail runners | 6 months
  The various repercussions listed in the questionnaires will be presented in terms of the percentage of women affected and their 95% confidence interval. The averages of the visual analog scale associated with their parameters of dispersion in order to evaluate the impact of SUI on everyday life and in their sporting activities will also be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bouscaren, MD, Principal Investigator — CHU La Réunion
Locations (1):
- CHU la Réunion, Saint-Denis, Reunion